CLINICAL TRIAL: NCT04905056
Title: A Prospective, Two-center, Single Arm Phase II Clinical Study to Evaluate Safety and Effectiveness of Ablation Therapy in the Treatment of Lung Cancer Presenting as Ground-glass Nodules
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Xi Junjie, professor, Shanghai Zhongshan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2021-088R
Record Dates: First submitted 2021-05-23; First posted 2021-05-27 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Progression
MeSH Terms: conditions — Disease Progression

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ablation therapy in the treatment of lung cancer presenting as ground-glass nodules (Experimental)
  Interventions: Other: Ablation therapy

INTERVENTIONS:
Other: Ablation therapy — Ablation therapy in the treatment of lung cancer presenting as ground-glass nodules

SUMMARY:
A prospective, two-center, single arm phase II clinical study to evaluate safety and effectiveness of ablation therapy in the treatment of lung cancer presenting as ground-glass nodules

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 85 years;
2. GGO is diagnosed by lung CT and failure to subside after 3 months (the patient having been re-examined by thin-section CT);
3. The maximum diameter of the GGO is bigger than 8mm and smaller than 3cm;
4. For single GGO: obvious progress was observed in pure GGO or the solid component of mixed ground glass nodules was more than or equal to 2 mm
5. The patients were unable to tolerate the operation for various reasons or multiple grinding glass nodules, operation can not be completely removed; or patients had received surgery in ipsilateral chest
6. The patient is able to understand and comply with the study and has provided written informed consent

Exclusion Criteria:

1. Patients who participated in any drug and / or medical device clinical trials within one month before the trial
2. had severe disease conditions
3. allergy to narcotic drugs
4. had other autoimmune disease
5. dementia or cognitive impairment can't cooperate with researchers
6. any local treatment other than ablation was received within 4 weeks before the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
progression free survival | 1 years
  One year progression free survival after radiofrequency ablation of ground glass nodules

SECONDARY OUTCOMES:
overall survival | 1 years, 3 years, 5years
  overall survival after radiofrequency ablation of ground glass nodules

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Thoracic Surgery, Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China